CLINICAL TRIAL: NCT01814150
Title: The Association Between Alpha 1 Acid Glycoprotein Level and Outcome of Patients With Metastatic Cancer Treated With Docetaxel Based Chemotherapy
Brief Title: The Association Between Alpha 1 Acid Glycoprotein Level and Outcome Metastatic Cancer Treated With Docetaxel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gottfried Maya (Other)
Responsible Party: Sponsor-Investigator, Gottfried Maya, Head, Institution of Oncology, Meir Medical Center
Organization: Meir Medical Center (Other)
Other Study IDs: A1AGP1234
Record Dates: First submitted 2013-03-05; First posted 2013-03-19 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Metastatic Lung Cancer; Metastatic Breast Cancer; Metastatic Gastric Cancer; Metastatic Prostate Cancer; Metastatic Bladder Cancer
Keywords: Docetaxel; Alpha 1 Acid Glycoprotein; Outcome
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Stomach Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oncology Institute, Meir Medical Center: Metastatic cancer patients treated with docetaxel at the Oncology Institute, Meir Medical Center

SUMMARY:
Docetaxel based chemotherapy is a standard therapy in various metastatic cancers including lung cancer, breast cancer, gastric cancer, prostate cancer, and bladder cancer.

One of the main plasma protein carriers of docetaxel is Alpha 1 acid glycoprotein.

Retrospective data suggests that plasma level of alpha 1 acid glycoprotein is associated with the outcome of docetaxel based therapy in cancer patients.

The investigators aim to prospectively study the association between the plasma level of alpha 1 acid glycoprotein and the outcome of docetaxel based therapy in cancer patients.

DETAILED DESCRIPTION:
Docetaxel based chemotherapy is a standard therapy in various metastatic cancers including non small cell lung cancer, breast cancer, gastric cancer, prostate cancer, and bladder cancer.

One of the main plasma protein carriers of docetaxel is Alpha 1 acid glycoprotein

Retrospective data suggests that plasma level of alpha 1 acid glycoprotein is associated with the outcome of docetaxel based therapy in non small cell lung cancer patients.

The investigators aim to prospectively study the association between the baseline plasma level of alpha 1 acid glycoprotein (measured on the first day of the first cycle of docetaxel) and the outcome (response rete, progression free survival, overall survival) of docetaxel based therapy in patients with metastatic non small cell lung cancer, breast cancer, stomach cancer, prostate cancer, and bladder cancer.

ELIGIBILITY:
Inclusion Criteria

* patients with metastatic cancer from lung, breast, gastric, prostate, and bladder origin
* patients must be treated with docetaxel based chemotherapy
* patients must sign an informed consent form

Exclusion Criteria

* patients with metastatic cancer other than lung, breast, gastric, prostate, and bladder origin
* patients treated with chemotherapy other than docetaxel
* patients that did not sign an informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Metastatic cancer from lung, breast, gastric, prostate, and bladder origin, treated with docetaxel based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
The association between the baseline plasma level of alpha 1 acid glycoprotein and progression free survival of docetaxel based therapy in patients with metastatic cancer | 3 years
  The association between the baseline plasma level of alpha 1 acid glycoprotein and progression free survival of docetaxel based therapy in patients with metastatic non small cell lung cancer, breast cancer, gastric cancer, prostate cancer, and bladder cancer

SECONDARY OUTCOMES:
The association between the baseline plasma level of alpha 1 acid glycoprotein and the response rate and overall survival of docetaxel based therapy in patients with metastatic cancer | 3 years
  The association between the baseline plasma level of alpha 1 acid glycoprotein and the response rate and overall survival of docetaxel based therapy in patients with metastatic non small cell lung cancer, breast cancer, gastric cancer, prostate cancer, and bladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Keizman, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Institute of Oncology, Meir Medical Center, Kfar Saba, Israel